CLINICAL TRIAL: NCT07119359
Title: Integrating HIV Prevention With TB Household Contact Evaluation in Uganda (TB PrEP)
Brief Title: Integrating HIV Prevention With TB Household Contact Evaluation in Uganda
Acronym: TB PrEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Ross, Assistant Professor, Department of Medicine, Division of Allergy and Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020907; R01MH134685 (NIH)
Record Dates: First submitted 2025-07-23; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis (TB); Human Immunodeficiency Virus (HIV) Prophylaxis
Keywords: Uganda; TB contact tracing; HIV; Tuberculosis; PrEP; Household
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Household randomized implementation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based HIV self-testing and PrEP initiation (Experimental): Home-based HIV self-testing and PrEP initiation (for eligible participants) integrated into routine TB household contact investigation
  Interventions: Other: Home-based HIV self-testing; Other: Home-based initiation of PrEP
- Modified standard of care (No Intervention): Referral to health facility for HIV testing and PrEP initiation

INTERVENTIONS:
Other: Home-based HIV self-testing — Integration of HIV self-testing into TB household contact investigation
  Arms: Home-based HIV self-testing and PrEP initiation
Other: Home-based initiation of PrEP — Integration of PrEP initation into TB household contact investigation
  Arms: Home-based HIV self-testing and PrEP initiation

SUMMARY:
This household randomized implementation study assesses the implementation and effectiveness of home-based HIV self- testing and PrEP initiation versus standard clinic referral for PrEP initiation during modified standard-of-care (modified SOC) household TB contact investigation in Uganda. It uses qualitative methods to evaluate the process of implementing the intervention and a health economic evaluation to assess the financial sustainability of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Person with pulmonary TB OR live in a household with someone with pulmonary TB being treated at one of the participating health facilities
* Household includes ≥2 persons
* Age 15 years and older
* Willingness to participate in study procedures

Exclusion Criteria:

* Lives in a congregate setting (e.g., dormitory or jail)
* Lives outside the study area
* Any other condition that, in the opinion of the Investigator/designee, could preclude informed consent, make study participation unsafe, or otherwise interfere with achieving study objectives

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2480 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | From enrollment to the one-month follow-up visit
  Uptake of PrEP among eligible household members, measured as the proportion initiating PrEP by 1 month and found to have detectable tenofovir use at the one-month visit

SECONDARY OUTCOMES:
PrEP continuation | From enrollment to six-month follow-up visit
  Proportion of participants initiating PrEP with detectable tenofovir in urine samples at three- and six-month visits
HIV testing coverage | From enrollment to six-month follow-up visit
  Proportion of participants known to be living with HIV or have tested HIV-negative among all participants

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Ross, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Select IPD will be available through the NIMH data archive
Access Criteria: Data will be shared through the NIMH Data Archive